CLINICAL TRIAL: NCT04964921
Title: Distinguishing Patient Groups Using Autonomic Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: DyAnsys, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CS011
Record Dates: First submitted 2021-07-03; First posted 2021-07-16 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Diabetes
Keywords: Impaired Fasting Glucose; Autonomic Dysfunction Measurement; Heart Rate Variability; Vital Signs Monitoring
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Impaired Fasting Glucose Individuals: The group contains subjects with various stages of impaired fasting glucose tolerance levels and diabetes (with or without complications). All subjects will be considered in one group since the heart rate variability and vital signs are monitored in a single visit.
  Interventions: Other: Device: ANSiScope Plus

INTERVENTIONS:
Other: Device: ANSiScope Plus — Heart rate variability measurement and vital signs monitoring will be performed on all subjects.

SUMMARY:
A study population with impaired fasting glucose levels, impaired glucose tolerance levels and diabetes (with or without complications) along with healthy patients will be chosen as participants. Their vital signs and their ECG (electrocardiograph) will be recorded during their only visit. Data analysis will be performed using the vital signs parameters. The RR intervals from the ECG will be analyzed by 5 different techniques to determine the best technique that stratifies the subjects the most accurately.

DETAILED DESCRIPTION:
The Autonomic Nervous System (ANS) is a fundamental part of the nervous system in the body. And yet, there is no technique to test or measure the health and functioning of a person's autonomic nervous system.This type of study will determine the most accurate methodology to test the autonomic nervous system through heart rate variability (HRV) monitoring and gain vital information to distinguish patient groups in the diabetic population.

There is no gold standard for measuring autonomic dysfunction. Currently the method of power spectral analysis is finding very wide usage. It Is known that power spectral analysis does not discriminate the two subsystems of the ANS well. There are other beat to beat methodologies that have not yet gained traction. The reason for conducting this trial is to take a group of subjects in various stages of impaired fasting glucose, impaired glucose tolerance and diabetes (with and without complications) and determine which methodology stratifies these subjects most accurately.

Our study aims to introduce a new measurement method named the 'Beat to Beat' (BB) method for gauging autonomic dysfunction in patients. The investigators hope to observe that the average beat to beat method (BB) score could help discriminating diabetic patients into the following five distinct groups from the pilot study:

1. Normal blood glucose level: - (A blood sugar level less than 140 mg/dL)
2. Impaired fasting glucose (IFG): - (A fasting blood sugar level from 100 to 125 mg/dL)
3. Impaired glucose tolerance (IGT): - (two-hour glucose levels of 140 to 199 mg per dL
4. Diabetes without complications: - (e.g., no neuropathy, no retinopathy or nephropathy)
5. Diabetes with complications: - (at least one complication among neuropathy, retinopathy, or nephropathy)

By showing that this measurement bears no relationship to the other four vital signs parameters (heart rate, blood oxygenation, blood pressure, body temperature), it will prove the necessity of this measurement in addition to the four vital signs for distinguishing patient groups among the diabetic population.

ELIGIBILITY:
Inclusion Criteria:

* Can provide informed consent.
* Age between 18 and 85 years old
* Body Mass Index: 25 ≤ BMI ≤ 40
* Hemoglobin A1c level: 7.5 ≤ HbA1c ≤ 9.5
* Individuals with pre-diabetes and diabetes Type II for at least 1 year (diagnosed by ADA criteria) and up to 20 years
* Advanced diabetic complications including neuropathy, nephropathy, retinopathy and other related complications
* Stable dose of medications for the previous 3 months
* Stable diet and lifestyle for the previous 3 months
* Stable medical status (Ex: no myocardial infarction, stroke, major surgery,

Exclusion Criteria:

* Unable to provide informed consent
* Chronic disease (e.g. HIV, Cushing syndrome, CKD, acromegaly, active hyperthyroidism etc.)
* Cancer and anticancer treatment in the last 5 years
* Psychiatric disorders (that in the eyes of the investigator should exclude the participant)
* Any disorder, which in the investigator's opinion might jeopardize subject's safety or compliance with the protocol
* Organ (kidney, pancreas, liver) transplant recipients
* Pregnancy or lactation
* Positive drug screen (opiates, methadone, cocaine, amphetamines, cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants and alcohol)
* Alcoholics or Smokers
* Positive screen on HBsAg, anti-HCV or anti-HIV ½
* History of diabetic ketoacidosis or hyperosmolar coma
* Subjects with known coronary artery disease or coronary revascularisation
* Subjects with previous history of cerebrovascular accident
* Subjects with known proliferative retinopathy or previous laser treatment for diabetic retinopathy
* Subjects with life-threatening conditions including malignancy
* Subjects with known psychiatric conditions including depression
* Subjects with significant renal impairment (eGFR<60ml/min at baseline) or non-diabetic renal disease (e.g. biopsy-proven glomerulonephritis or obstructive uropathy)
* Subjects with major physical disability

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults of either sex with various stages of impaired fasting glucose tolerance levels and diabetes (with or without complications) will be considered as study population.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Determination of autonomic dysfunction by subject | The measurement will happen in a single visit i.e 1 day.
  The ANSiScope Plus will be used to determine the BB (beat to beat) score through heart rate variability measurements.

SECONDARY OUTCOMES:
Establish the absence of any relationship of autonomic dysfunction (AD) to any other vital signs parameters. | The measurement will happen in a single visit i.e 1 day.
  Investigate the importance of measuring the autonomic dysfunction in the presence of other vital signs measurements (heart rate, body temperature, blood oxygenation and blood pressure)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Bathula Sridhar, MD,DM (Endo), Principal Investigator — Samraksha Diabetes, Thyroid, Endocrine Superspecialty Hospital and Research Centre